CLINICAL TRIAL: NCT00316654
Title: A Phase IV,Multi-Center,Open-Label,Unrandomized Study to Evaluate the Persistence of Antibody Response to N.Meningitidis Group C,Before & After 2 Doses of the Conjugate Pneumococcal Vaccine,in Children Seven Months & Older Who Previously Received Immunization With Chiron Meningococcal C Conjugate Vaccine & a Hexavalent Infant Vaccine According to the Applicable Infant Immunization Schedule
Brief Title: Persistence of Antibody Response to N. Meningitidis Group C in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V14P38E1; 2004-001522-24 (EudraCT Number)
Record Dates: First submitted 2006-04-19; First posted 2006-04-21 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Prevention of Meningococcal Infection
Keywords: Prevention of Meningococcal Meningitis; vaccines, conjugate; immunology; child; antibody persistence
MeSH Terms: interventions — serogroup C meningococcal conjugate vaccine

INTERVENTIONS:
Biological: Meningococcal C conjugate vaccine

SUMMARY:
Persistence of Antibody Response to N. meningitidis Group C in Children

ELIGIBILITY:
Inclusion Criteria:

* healthy children

Exclusion Criteria:

* previous ascertained or suspected disease caused by N. meningitidis
* previous significant acute or chronic infections
* any other serious disease

Min Age: 7 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 489 (Actual)
Dates: Start 2005-02; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Immunogenicity: serum antibody responses, as measured by bactericidal activity,using hBCA

SECONDARY OUTCOMES:
Evaluate and compare persistence of antibody response to N. meningitidis serogroup C as measured by serum bactericidal activity
safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines Drug Information Services, Principal Investigator — Novartis Vaccines & Diagnostics
Locations (2):
- Olsztyn, Lubartów, Kielce, Kraków, Bydgoszcz, Poland
- Valencia, Spain